CLINICAL TRIAL: NCT05694598
Title: A Phase 1 Study to Assess the Safety and Tolerability of VGR-R01 in Patients With Bietti Crystalline Dystrophy
Brief Title: Safety and Tolerability of VGR-R01 for Patients With Bietti Crystalline Dystrophy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGR-R01-101
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bietti Crystalline Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGR-R01 (Experimental): Single-dose Subretinal Administration of VGR-R01
  Interventions: Genetic: VGR-R01

INTERVENTIONS:
Genetic: VGR-R01 — CYP4v2-coding gene delivered by AAV vector

SUMMARY:
A Multicenter, Open-Label, Non-Randomized, Uncontrolled Study of VGR-R01 in Patients with Bietti Crystalline Dystrophy.

DETAILED DESCRIPTION:
VGR-R01 is a novel AAV vector carrying the human CYP4V2 coding sequence. This study is intended to evaluate the safety and tolerability of a single subretinal administration of VGR-R01. All subjects will undergo at least 52 weeks of safety observation and will be encouraged to enroll in an extension study to evaluate the long-term safety of VGR-R01 for a total of five years.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to provide informed consent and comply with requirements of the study;
2. ≥18 years and <70 years of age;
3. Confirmed diagnosis of Bietti Crystalline Dystrophy and molecular diagnosis of CYP4V2 mutations (homozygotes or compound heterozygotes);
4. BCVA ≤ 60 ETDRS letters in the study eye.

Key Exclusion Criteria:

1. Have insufficient viable retinal photoreceptor cells based on investigator's decision;
2. Have current ocular or periocular infections, or endophthalmitis;
3. Have any significant ocular disease/disorder other than BCD, including age-related macular degeneration, diabetic retinopathy, optic neuropathy, significant lens opacity, glaucoma, uveitis, retinal detachment, etc;
4. Have intraocular surgery history except cataract surgery in the study eye;
5. Have or potentially require of systemic medications that may cause eye injure;
6. Have contraindications for corticosteroids or immunosuppressant;
7. Unwilling or unable to have the planned follow-up;
8. Abnormal coagulation function or other clinically significant abnormal laboratory results;
9. Have malignancies or history of malignancies;
10. History of immunodeficiency (acquired or congenital); Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2028-09-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Baseline up to Week 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of serious adverse events | Baseline up to Week 52
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that resulted in death; life threatening; require inpatient hospitalization or prolongation of existing hospitalization; result in persistent or significant disability/incapacity; result in congenital anomaly/birth defect.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs | Baseline up to Week 52
  Vital signs (temperature, respiratory rate, pulse rate, systolic and diastolic blood pressure) will be obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs will be determined at the investigator's discretion.
Number of Participants with Clinically Laboratory Abnormalities | Baseline up to Week 52
  Laboratory Tests will include hematology, coagulation, blood chemistry, urinalysis, serology, and pregnancy test, etc. If any potential changes accompanied by clinical symptoms, or results in a change of medical intervention, the findings will be considered as clinically significant based on investigator's decision.
Number of Participants with Clinically Significant Change from Baseline in Ophthalmic Examination Findings | Baseline up to Week 52
  Ophthalmic Examination will include BCVA, IOP, slitlamp examination, angiography and SD-OCT, etc. If any potential changes accompanied by clinical symptoms, or results in a change of medical intervention, the findings will be considered as clinically significant based on investigator's decision.

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | Week 52
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured.
Changes from baseline of Visual Field Index (%) in Visual Field (Humphery perimetry) indexes | Week 52
  The VFI can range from 100% (normal visual field) to 0% (perimetrically blind field).
Changes from baseline of Mean Deviation (dB) in Visual Field (Humphery perimetry) indexes | Week 52
  Normal values are typically within 0dB and -2dB.
Changes from baseline of Pattern Standard Deviation (dB) in Visual Field (Humphery perimetry) indexes | Week 52
  A typical "normal" dB reading is around 30. The numeric dB graph should be studied next. The dBs tested by the Humphrey analyzer range between 0 and 50 dB (0 is the brightest and 50 is the dimmest).
Changes from baseline in Mobility testing scores | Week 52
  The mobility score range is between -1 (the worst functional vision) and 6 (the best).

OTHER OUTCOMES:
Patient reported outcome: Changes of NEI-VFQ-25 | Week 52
  NEI-VFQ-25 questionnaire measures dimensions of self-reported vision-targeted health status that are most important to persons with eye disease. Total score ranges from 0-100, where a score of 0 represents the worst outcome and 100 represents the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Shanghai Vitalgen Biopharma Co.,Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGR-R01 is fully approved.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be shared with other researchers when VGR-R01 is fully approved.
Access Criteria: IPD will be shared with other researchers when VGR-R01 is fully approved.